CLINICAL TRIAL: NCT03980925
Title: A Phase II Study of Platinum-doublet Chemotherapy in Combination With Nivolumab as First-line Treatment in Subjects With Unresectable, Locally Advanced or Metastatic G3 Neuroendocrine Neoplasms (NENs) of the Gastroenteropancreatic (GEP) Tract or of Unknown (UK) Origin.
Brief Title: Platinum-doublet Chemotherapy and Nivolumab for the Treatment of Subjects With Neuroendocrine Neoplasms (NENs) of the Gastroenteropancreatic (GEP) Tract or of Unknown (UK) Origin.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-T1913
Record Dates: First submitted 2019-06-07; First posted 2019-06-10 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Neoplasm; Gastroenteropancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Gastro-enteropancreatic neuroendocrine tumor | interventions — Nivolumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab + platinum-doublet chemotherapy (Experimental): 1. Induction Phase: Nivolumab 360 mg IV plus Carboplatin IV (AUC=5) plus Etoposide 10mg/m2/day on days 1-3D, all every 3 weeks up to 6 cycles followed by Nivolumab 480mg for 24 months or until progression of the disease (PD), death or toxicity.
     Order of administration: Nivolumab, Carboplatin, Etoposide
  2. Maintenance Phase Nivolumab 480 mg IV will be administered every 4 weeks (±3 days) for 2 years.
  Interventions: Drug: Nivolumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Nivolumab — Subjects will receive Nivolumab 360 mg every 3 weeks (Q3W) first day of each cycle plus Carboplatin area under the curve (AUC5) Q3W first day of each cycle plus Etoposide 100 day 1-3 of each cycle up to 6 cycles of combined therapy (Induction Phase).
  At the time of completion of 6 cycles of chemotherapy and nivolumab, participants who have not experienced disease progression will continue to receive nivolumab at a dose of 480 mg as 30 minute infusion every 4 weeks for up to 2 years (24 months) (maintenance phase).
  Cycles are defined by 4 weeks or 28 days.
Drug: Carboplatin — Subjects will receive Nivolumab 360 mg every 3 weeks (Q3W) first day of each cycle plus Carboplatin AUC5 Q3W first day of each cycle plus Etoposide 100 day 1-3 of each cycle up to 6 cycles of combined therapy (Induction Phase).
  At the time of completion of 6 cycles of chemotherapy and nivolumab, participants who have not experienced disease progression will continue to receive nivolumab at a dose of 480 mg as 30 minute infusion every 4 weeks for up to 2 years (24 months) (maintenance phase).
  Cycles are defined by 4 weeks or 28 days.
Drug: Etoposide — Subjects will receive Nivolumab 360 mg every 3 weeks (Q3W) first day of each cycle plus Carboplatin AUC5 Q3W first day of each cycle plus Etoposide 100 day 1-3 of each cycle up to 6 cycles of combined therapy (Induction Phase).
  At the time of completion of 6 cycles of chemotherapy and nivolumab, participants who have not experienced disease progression will continue to receive nivolumab at a dose of 480 mg as 30 minute infusion every 4 weeks for up to 2 years (24 months) (maintenance phase).
  Cycles are defined by 4 weeks or 28 days.

SUMMARY:
This is a prospective, multi-centre, open label, non-randomized phase II study evaluating the efficacy and safety of nivolumab plus platinum-based chemotherapy in patients with advanced G3 NENs of the GEP tract or of UK origin.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed G3 NENs originated in the gastroenteropancreatic tract (WHO 2010 classification). Patients with a G3 NEN of unknown primary will also be eligible for this trial.
* Ki-67 >20% or mitotic rate > 20 per 10 High-power field (HPF).
* Metastatic or locally advanced unresectable disease not amenable to treatment with curative intent.
* No prior systemic treatment for advanced disease nor as adjuvant therapy.
* Availability of fresh or archive formalin-fixed, paraffin-embedded tumor tissue for biomarker assessment.
* Patients must have clinically and/or radiographically documented measurable disease. At least one site of disease must be unidimensionally measurable as per RECIST 1.1.
* Adequate organ function as defined by the following criteria (within 7 days prior to enrollment):

  1. absolute neutrophil count (ANC) ≥1500 cells/mm3
  2. platelets ≥100,000 cells/mm3
  3. hemoglobin ≥9.0 g/dL
  4. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN); in patients with liver metastases AST and ALT ≤5.0 x ULN
  5. total bilirubin ≤1.5 x ULN
  6. serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥60 mL/min.
* Male or female, age ≥18 years.
* Eastern cooperative oncology group (ECOG) performance status of 0-2.
* Life expectancy of ≥12 weeks.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to treatment initiation.
* Highly effective contraception (i.e. methods with a failure rate of less than 1 % per year) for both fertile, sexually active male and female subjects. Highly effective contraception must be used 28 days prior to first trial treatment administration, for the duration of trial treatment, and at least for 60 days after stopping trial treatment.
* Signed and dated informed consent document must be given according to international conference harmonisation (ICH)/ Good clinical practice (GCP), and national/local regulations indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrolment.

Exclusion Criteria:

* The following endocrine tumor types may not be included: paraganglioma, adrenal, thyroid parathyroid or pituitary endocrine tumors. Large or small cell lung neuroendocrine carcinoma of the lung will also be excluded.
* Prior therapy with any immune checkpoint inhibitor.
* Major surgery, except diagnostic biopsy, in <4 weeks or radiation therapy <2 weeks prior to starting study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* Prior organ transplantation, including allogeneic stem-cell transplantation.
* Prior history of non-infectious pneumonitis requiring steroids or current pneumonitis.
* Systemic chronic steroid therapy (> 10 mg/day prednisone or equivalent) or other immunosuppressive agents or use of any investigational drug within 28 days before the start of trial treatment. Short-term administration of steroids for allergic reactions or management of immune-related adverse events is allowed. Topical, inhaled, nasal and ophthalmic steroids are also allowed.
* Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment.
* Known history of positive testing for Human Immunodeficiency Virus (HIV) infection, known history of or positive tests for Hepatitis B virus surface antigen (HBVsAg) or Hepatitis C ribonucleic acid (HCV RNA) indicating acute or chronic infection or other significant acute or chronic infections requiring medication at study entry.
* Active, known or suspected autoimmune disease or a documented history of autoimmune disease, including ulcerative colitis and Crohn's disease. (Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll).
* Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment will not be allowed to enter the study. Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, new york heart association (NYHA) class > III congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism.
* Known hypersensitivity reactions to monoclonal antibodies (≥ grade 3 according to NCI Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 [xliii] or any past medical history of anaphylaxis or uncontrolled asthma (i.e., 3 or more asthma characteristics partially controlled).
* Any other prior malignancy within 5 years of study entry, with the exception of adequately treated in-situ carcinoma of the cervix, breast or uteri, or non-melanomatous skin cancer.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Female patients who are pregnant or lactating, or men and women of reproductive potential not willing or not able to employ an effective method of birth control/contraception to prevent pregnancy during treatment and for 6 months after discontinuing study treatment The definition of effective contraception should be in agreement with local regulation and based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rocío García-Carbonero, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre; Maria del Carmen Riesco-Martínez, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre
Locations (12):
- Spain (12):
  - Institut Català d'Oncologia Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson Cancer Madrid, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + Platinum-doublet Chemotherapy: 1. Induction Phase: Nivolumab 360 mg IV plus Carboplatin IV (AUC=5) plus Etoposide 10mg/m2/day on days 1-3D, all every 3 weeks up to 6 cycles followed by Nivolumab 480mg for 24 months or until PD, death or toxicity.
     Order of administration: Nivolumab, Carboplatin, Etoposide
  2. Maintenance Phase Nivolumab 480 mg IV will be administered every 4 weeks (±3 days) for 2 years.
Period: Induction Phase
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Started | 37
Completed | 37
Not Completed | 0
Period: Maintenance Phase
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Combination of Nivolumab and Platinum-doublet Chemotherapy: Patients with unresectable advanced or metastatic G3 (Ki-67 >20% or mitotic rate >20 per 10 high-power fields (HPF) neuroendocrine neoplasms (NENs) of gastroenteropancreatic (GEP) or unknown origin treated with a combination of nivolumab and platinum-doublet chemotherapy.
Arm/Group | Combination of Nivolumab and Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 61.0 [28 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 34
  Latin | 2
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  Spain | 37
ECOG [Count of Participants; unit: Participants] — The ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 (Fully active, able to carry on all pre-disease performance without restriction) to 5 (Dead).
  Participants
    0 | 11
    1 | 22
    2 | 4
Stage at diagnosis [Count of Participants; unit: Participants]
  I | 1
  III | 1
  IV | 35
Differentiation [Count of Participants; unit: Participants]
  Neuroendocrine tumor (NET) | 12
  Neuroendocrine carcinoma (NEC) | 25
Ki-67 [Count of Participants; unit: Participants] — KI-67 antigen is a nuclear protein associated with cell proliferation. It is a cellular marker of proliferation that can be used in immunohistochemistry. The percentage of cells in the field that have positive expression/presence of KI-67 is reported here. A higher percentage indicates greater proliferation, more aggressive tumor.
  Participants
    21 - 55% | 12
    >55% | 25
Primary site [Count of Participants; unit: Participants]
  Esophageal | 2
  Gastric | 6
  Pancreatic | 14
  Colonic | 4
  Rectal | 2
  Small intestine | 2
  Other | 2
  Unknown | 5
Metastatic sites number [Count of Participants; unit: Participants]
  1 | 10
  ≥2 | 27
Metastasis sites [Count of Participants; unit: Participants]
  Liver | 31
  Lung | 9
  Lymph nodes | 18
  Bone | 10
Previous surgery [Count of Participants; unit: Participants]
  Yes | 6
  No | 30
  Unknown | 1
Cromogranin A (CgA) [Count of Participants; unit: Participants]
  < 2x upper limit normal (ULN) | 7
  ≥ 2x ULN | 27
  Unknown | 3
Enolase [Count of Participants; unit: Participants]
  < 2x ULN | 13
  ≥ 2x ULN | 21
  Unknown | 3
Lactate dehydrogenase (LDH) [Count of Participants; unit: Participants]
  > 2x ULN | 9
  ≤ 2x ULN | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 12 Months
Description: Percentage of patients alive at 1-year from first dose of treatment.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
% of participants | 54.1 [40.2 to 72.8]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Response to treatment according to RECIST 1.1 criteria or iRECIST 1.1 criteria assessed by computed tomography (CT) scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Throughout the study period, approximately 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
percentage of participants | 56.8

3. Secondary Outcome: Progression-free Survival (PFS) Rate
Description: Percentage of patients without progression of disease (PD) calculated from the date of treatment initiation with first-line chemotherapy and nivolumab until the date of first documentation of PD as per RECIST v1.1 or death.
Time Frame: Throughout the study period, approximately 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
percentage of participants
  PFS at 12 months | 21.6 [11.7 to 39.9]
  PFS at 24 months | 8.1 [2.7 to 24]

4. Secondary Outcome: Median Overall Survival
Description: Length of time between start of treatment and death
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
months | 13.9 [8.3 to 30]

5. Secondary Outcome: Predictive Biomarkers
Description: Assess biochemical response in patients with baseline elevation of enolase and correlate it with clinical outcome.
Time Frame: 30 months
Measure: Number; unit: Percentage of patients with response
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
Percentage of patients with response | 52.4

6. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Number and type of adverse events reported throughout the study period according to CTCAE 5.0 criteria.
Time Frame: 30 months
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
percentage of participants
  Fatigue | 60.5
  Neutropenia | 55.3
  Nausea | 44.7
  Anemia | 31.6
  Alopecia | 31.6
  Diarrhea | 29
  Vomiting | 21.1
  Thrombopenia | 21.1
  Anorexia | 18.4
  Mucositis | 15.8

7. Secondary Outcome: Median Progression-free Survival
Description: Length of time between date of evidenced response and progression of disease or death
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
months | 5.7 [5.1 to 9]

8. Secondary Outcome: Duration of Response
Description: The percentage of patients achieving Complete Response, Partial Response or stable disease (SD)
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
Number analyzed (Participants) | 37
month | 6.4 [3.2 to 11.1]

ADVERSE EVENTS:
Time Frame: 30 months
Description: Safety data was closely monitored by the contract research organization (CRO) with real time review and assesment of serious adverse events (SAEs) as they were received, and periodic review of all adverse events data for potential new safety signals.
Arm/Group | Nivolumab + Platinum-doublet Chemotherapy
All-Cause Mortality (participants affected / at risk) | 25/37
Serious Adverse Events (participants affected / at risk) | 18/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Platinum-doublet Chemotherapy (N=37)
Bowel subocclusion (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Platelet count decreased (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Immune-mediated nephritis (Renal and urinary disorders) | 1
Covid-19 (Infections and infestations) | 4
Acute kidney injury (Injury, poisoning and procedural complications) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Fever (General disorders) | 1
Inguinal hernia (Surgical and medical procedures) | 1
Sepsis (Infections and infestations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bacteremia (Infections and infestations) | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Esophageal mucositis (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
General clinical deterioration (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Confusion (Psychiatric disorders) | 1
Dysarthria (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Hepatic infection (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Platinum-doublet Chemotherapy (N=37)
Fatigue (General disorders) | 29
Neutrophil count decreased (Blood and lymphatic system disorders) | 21
Nausea (Gastrointestinal disorders) | 19
Anemia (Blood and lymphatic system disorders) | 18
Diarrhea (Gastrointestinal disorders) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 12
Vomiting (Gastrointestinal disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 10
Platelet count decreased (Blood and lymphatic system disorders) | 9
Gastrointestinal disorders (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 9
Fever (General disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 4
General disorders and administration site conditions (General disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Edema limbs (General disorders) | 4
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Hepatobiliary disorders (Hepatobiliary disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
White blood cell decreased (Blood and lymphatic system disorders) | 3
Endocrine disorders (Endocrine disorders) | 3
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pain (General disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Alanine aminotransferase increased (Investigations) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Aspartate aminotransferase increased (Investigations) | 2
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3
Headache (Nervous system disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Hyperthyroidism (Endocrine disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal and urinary disorders (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03980925/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03980925/SAP_001.pdf